CLINICAL TRIAL: NCT01225822
Title: BIBR 1048 Dose Range Finding Study in Prevention of Venous Thromboembolism in Patients With Primary Elective Total Hip or Knee Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1160.19
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Results first posted 2010-12-16 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-02

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin; Dabigatran

ARMS (5):
- BIBR 1048 50 mg bis in die(b.i.d) (Experimental): BIBR 1048 50 mg b.i.d twice a day plus two capsules of placebo matching BIBR 1048 0 mg twice a day plus one placebo matching enoxaparin 0 mg once a day for the treatment period
  Interventions: Drug: BIBR 1048
- BIBR 1048 150 mg b.i.d (Experimental): BIBR 1048 150 mg b.i.d twice a day plus two capsules of placebo matching BIBR 1048 0 mg twice a day plus placebo matching enoxaparin 0 mg once a day for the treatment period
  Interventions: Drug: BIBR 1048
- BIBR 1048 225 mg b.i.d (Experimental): BIBR 1048 225 mg b.i.d twice a day plus two capsules of placebo matching BIBR 1048 0 mg twice a day plus placebo matching enoxaparin 0 mg once a day for the treatment period
  Interventions: Drug: BIBR 1048
- BIBR 1048 300 mg quaque die(q.d) (Experimental): BIBR 1048 150 mg q.d once a day plus placebo matching BIBR 1048 0 mg twice a day plus placebo matching enoxaparin 0 mg once a day for the treatment period
  Interventions: Drug: BIBR 1048
- Enoxaparin 40 mg subcutaneous(s.c) (Active Comparator): placebo matching BIBR 1048 0 mg twice a day plus enoxaparin 40 mg s.c once a day for the treatment period
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Enoxaparin 40 mg s.c once a day for 5-10 days of treatment period
  Arms: Enoxaparin 40 mg subcutaneous(s.c)
Drug: BIBR 1048 — 50 mg b.i.d BIBR 1048 capsule twice a day for 5-10 days of treatment period
  Arms: BIBR 1048 50 mg bis in die(b.i.d)
Drug: BIBR 1048 — 150 mg b.i.d BIBR 1048 capsule twice a day for 5-10 treatment period
  Arms: BIBR 1048 150 mg b.i.d
Drug: BIBR 1048 — 225 mg b.i.d BIBR 1048 capsule twice a day for 5-10 treatment period
  Arms: BIBR 1048 225 mg b.i.d
Drug: BIBR 1048 — 300 mg q.d BIBR 1048 capsule for 5-10 treatment period
  Arms: BIBR 1048 300 mg quaque die(q.d)

SUMMARY:
The primary objective of this study is to establish the dose-response relationship with regard to efficacy and safety of BIBR 1048 (50 mg bis in die(b.i.d), 150 mg b.i.d, 225 mg b.i.d. and 300 mg quaque die(q.d) ) in preventing venous thromboembolism(VTE) in patients undergoing primary elective total hip and knee replacement.

ELIGIBILITY:
Inclusion criteria

1. Patients scheduled to undergo a primary elective total hip or knee replacement.
2. Male of female being 18 years or older.
3. Patients weighing at least 40 kg.
4. Written informed consent for study participation.

Exclusion criteria

1. Bleeding diathesis, constitutional or acquired coagulation disorders.
2. Major surgery or trauma(e.g., hip fracture) within the last 3 months.
3. Cardiovascular disease
4. Any history of haemorrhagic stroke, intracranial or intraocular bleeding or cerebral ischaemic attacks lasting more than 24 hours and / or with cardiovascular pathological findings.
5. Deep vein thrombosis(DVT), gastrointestinal or pulmonary bleeding, gastric or duodenal ulcer within the last year.
6. History of or acute intracranial disease
7. Liver disease
8. Renal disease
9. Use of long-term anticoagulants or antiplatelet drugs within 7 days prior to hip/knee replacement operation.
10. Pre-menopausal women who are not surgically steriles, are nursing and are of child-bearing potential and are not practising acceptable methods of birth control
11. Known allergy to contrast media
12. Thrombocytopenia
13. Allergy against heparin.
14. Active malignant disease or current cytostatic treatment.
15. Treatment with an investigational drug in the past month.
16. Leg amputee
17. Known alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1973 (Actual)
Dates: Start 2002-11; Primary Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (59):
- Austria (3):
  - 1160.19.43004 Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - 1160.19.43002 Orthopädisches Spital Speising, Vienna
  - 1160.19.43001 A.ö. Krankenhaus d. Statutarstadt Wiener Neustadt, Wiener Neustadt
- Belgium (5):
  - 1160.19.32002 V.U.B. Jette, Brussels
  - 1160.19.32004 UZ Gent, Ghent
  - 1160.19.32005 Virga Jesseziekenhuis, Ghent
  - 1160.19.32006 Boehringer Ingelheim Investigational Site, Huy
  - 1160.19.32007 C.H.U. de Tivoli, La Louvière
- Czechia (6):
  - 1160.19.42004 University Hospital Brno, Brno-Bohunice
  - 1160.19.42001 Hospital Kladno, Kladno
  - 1160.19.42006 Hospital Mlada Boleslav, Mladá Boleslav
  - 1160.19.42003 University Hospital Ostrava, Ostrava
  - 1160.19.42005 University Hospital Plzen, Pilsen
  - 1160.19.42009 University Hospital Na Bulovce, Prague
- Denmark (5):
  - 1160.19.45042 Orthopedic Surgical Clinic, Frederiksberg
  - 1160.19.45045 Gentofte Hospital, Hellerup
  - 1160.19.45043 Herlev Hospital, Herlev
  - 1160.19.45041 Hørsholm Sygehus, Hørsholm
  - 1160.19.45044 Orthopedic Surgical Dept., Silkeborg
- Finland (2):
  - 1160.19.35802 Keski-Suomen keskussairaala, Jyväskylä
  - 1160.19.35801 Oulun yliopistollinen sairaala, Leikkaus- ja tehohoidon yks., Oulu
- France (5):
  - 1160.19.33004 Div, Illkirch-Graffenstaden
  - 1160.19.33007 Clinique du Mail, La Rochelle
  - 1160.19.33009 Hôpital Edouard Herriot, Lyon
  - 1160.19.33006 Clinique Mutualiste, Saint-Etienne
  - 1160.19.33008 Clinique de l'Atlantique, Saint-Herblain
- Hungary (5):
  - 1160.19.36003 Sándor Péterfy Hospital, Budapest
  - 1160.19.36001 Kálmán Pándy County Hospital, Gyula
  - 1160.19.36004 Bács-Kiskun County Hospital, Kecskemét
  - 1160.19.36002 Albert Szent-Györgyi Medical and Pharmacological Center, Szeged
  - 1160.19.36005 Szent György Hospital, Székesfehérvár
- Italy (5):
  - 1160.19.39003 U. O. Ortopedia e Traumatologia, Bergamo
  - 1160.19.39005 Modulo Coordinazione Dipartimentale di Ricerca e Anestesia, Bologna
  - 1160.19.39002 Fondazione Centro S. Raffaele, Milan
  - 1160.19.39001 IRCCS Policlinico San Matteo, Pavia
  - 1160.19.39004 Ospedale di Circolo di Varese, Varese
- Netherlands (5):
  - 1160.19.31001 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.19.31003 Boehringer Ingelheim Investigational Site, Hilversum
  - 1160.19.31005 Hengstdal 3, Nijmegen
  - 1160.19.31006 Boehringer Ingelheim Investigational Site, Sittard
  - 1160.19.31004 Boehringer Ingelheim Investigational Site, Zwolle
- Norway (7):
  - 1160.19.47003 Helse Sunnmøre HF, Ålesund sykehus, Ålesund
  - 1160.19.47001 Nordlandssykehuset HF, Bodø, Bodø
  - 1160.19.47004 Martina Hansens Hospital, Bærum Postterminal
  - 1160.19.47008 Martina Hansens Hospital, Bærum Postterminal
  - 1160.19.47007 Sykehuset Innlandet HF, Avd. Elverum, Elverum
  - 1160.19.47005 Haugesund sjukehus HF, Haugesund
  - 1160.19.47002 Sykehuset Telemark HF, Avd. Skien, Skien
- South Africa (2):
  - 1160.19.27001 Dept. of Haematology, Johannesburg
  - 1160.19.27002 Suite 203, Johannesburg
- Sweden (9):
  - 1160.19.46002 Kirurgavdelningen, Falköping
  - 1160.19.46001, Gothenburg
  - 1160.19.46004 Ortopediska kliniken, Länssjukhuset, Halmstad, Halmstad
  - 1160.19.46003 Ortopediska kliniken, Länssjukhuset i Kalmar, Kalmar
  - 1160.19.46007 Kungälvs sjukhus, Kungälvs
  - 1160.19.46005 Kirurg Ortopediska kliniken, Sjukhuset i Lidköping, Lidköping
  - 1160.19.46008 Ortopediska Institutionen, Linköping
  - 1160.19.46009 Sahlgrenska Universitetssjukhuset, Mölndal, Mölndal
  - 1160.19.46006 Boehringer Ingelheim Investigational Site, Varberg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 1973 patients enrolled/randomised in this trial but only 1949 started treatment
Groups:
- BIBR 1048 50 mg Bid: Dabigatran 50 mg bid(twice daily) oral
- BIBR 1048 150 mg Bid: Dabigatran 150 mg bid(twice daily) oral
- BIBR 1048 225 mg Bid: Dabigatran 225 mg bid(twice daily) oral
- BIBR 1048 300 mg qd: Dabigatran 300 mg qd(once daily) oral
- Enoxaparin 40 mg qd: Enoxaparin 40 qd (once daily) subcutaneous injection
Period: Overall Study
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Started | 389 | 390 | 393 | 385 | 392
Completed | 351 | 334 | 355 | 333 | 361
Not Completed | 38 | 56 | 38 | 52 | 31
Not completed — Adverse Event | 13 | 31 | 18 | 23 | 14
Not completed — Protocol Violation | 6 | 8 | 6 | 7 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 7 | 7 | 11 | 6
Not completed — Other | 13 | 10 | 7 | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- BIBR 1048 50 mg Bid: Dabigatran 50 mg bid (twice daily) oral
- BIBR 1048 150 mg Bid: Dabigatran 150 mg bid (twice daily) oral
- BIBR 1048 225 mg Bid: Dabigatran 225 mg bid (twice daily) oral
- BIBR 1048 300 mg qd: Dabigatran 300 mg qd (once daily) oral
- Enoxaparin 40 mg qd: Enoxaparin 40 mg qd (once daily) subcutaneous injection
- Total: Total of all reporting groups
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd | Total
Number analyzed (Participants) | 389 | 390 | 393 | 385 | 392 | 1949
Age, Customized [Mean (Standard Deviation); unit: years] — Safety set population
  years | 66.07 (10.23) | 65.86 (10.77) | 65.87 (10.63) | 66.47 (10.37) | 65.03 (11.03) | 65.86 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety set population
  Participants
    Female | 223 | 252 | 229 | 246 | 241 | 1191
    Male | 166 | 138 | 164 | 139 | 151 | 758

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Venous Thromboembolic (VTE) Events
Description: Deep vein thrombosis (DVT) (proximal and distal) as detected by routine bilateral venography on day 8 +/- 2, plus symptomatic DVT confirmed by venography during the treatment period or PE confirmed by objective testing
Time Frame: Treatment period (up to day 8+/-2 days visit)
Population: Full Analysis Set (FAS) population. This included all randomised patients who had at least one subcutaneous injection and one oral dose of study medication and with confirmed VTE data post surgery
Measure: Number; unit: participants
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 372 | 375 | 381 | 371 | 382
participants | 86 | 49 | 39 | 47 | 72
Statistical Analysis 1: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 225 mg Bid; BIBR 1048 225 mg bid vs. BIBR 1048 50 mg bid comparison. The primary objective of the trial was to establish a dose relationship among BIBR 1048 doses studied in the prevention of VTE. The statistical model was a logistic regression which included treatment and centre; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Dose relationship tested using a hierarchical testing procedure to preserve type I error rate at 5%. 225 mg bid was compared to 50 mg bid. If a difference significant at 5% level was found, then 150 mg bid was compared to 50 mg bid; Odds Ratio (OR) = 0.375, 95% CI [0.244 to 0.577]
Statistical Analysis 2: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 150 mg Bid; BIBR 1048 150 mg bid vs. BIBR 1048 50 mg bid comparison. The primary objective of the trial was to establish a dose relationship among BIBR 1048 doses studied in the prevention of VTE. The statistical model was a logistic regression which included treatment and centre; Test type: Superiority or Other; p = 0.0015, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.518, 95% CI [0.344 to 0.778]
Statistical Analysis 3: Comparison: BIBR 1048 150 mg Bid vs BIBR 1048 300 mg qd; BIBR 1048 300 mg qd vs. BIBR 1048 150 mg bid comparison. Secondary analysis to compare once daily dosing vs. twice daily dosing. . The statistical model was a logistic regression which included treatment and centre; Test type: Superiority or Other; p = 0.7856, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI [0.599 to 1.473]
Statistical Analysis 4: Comparison: BIBR 1048 225 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 225 mg bid vs. Enoxaparin 40 mg qd comparison. Secondary analysis, active control used as reference. The statistical model was a logistic regression which included treatment and centre; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 0.469, 95% CI [0.302 to 0.727]
Statistical Analysis 5: Comparison: BIBR 1048 150 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 150 mg bid vs. Enoxaparin 40 mg qd comparison. Secondary analysis, active control used as reference. The statistical model was a logistic regression which included treatment and centre; Test type: Superiority or Other; p = 0.0401, Regression, Logistic; Odds Ratio (OR) = 0.647, 95% CI [0.427 to 0.98]
Statistical Analysis 6: Comparison: BIBR 1048 50 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 50 mg bid vs. Enoxaparin 40 mg qd comparison. Secondary analysis, active control used as reference. The statistical model was a logistic regression which included treatment and centre; Test type: Superiority or Other; p = 0.2446, Regression, Logistic; Odds Ratio (OR) = 1.249, 95% CI [0.859 to 1.817]

2. Secondary Outcome: Number of Participants With VTE Events and All Cause Mortality
Description: Deep venous thrombosis (DVT) (proximal and distal) as detected by routine bilateral venography on day 8 +/- 2, plus symptomatic DVT confirmed by venography during the treatment period or Pulmonary Embolism (PE) confirmed by objective testing and all deaths.
Time Frame: Treatment period (up to day 8+/-2 days visit)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 372 | 375 | 381 | 371 | 382
participants | 86 | 49 | 39 | 47 | 72
Statistical Analysis 1: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 225 mg Bid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.375, 95% CI [0.244 to 0.577]
Statistical Analysis 2: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 150 mg Bid; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0015, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.518, 95% CI [0.344 to 0.778]
Statistical Analysis 3: Comparison: BIBR 1048 150 mg Bid vs BIBR 1048 300 mg qd; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.7856, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI [0.599 to 1.473]
Statistical Analysis 4: Comparison: BIBR 1048 225 mg Bid vs Enoxaparin 40 mg qd; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 0.469, 95% CI [0.302 to 0.727]
Statistical Analysis 5: Comparison: BIBR 1048 150 mg Bid vs Enoxaparin 40 mg qd; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.0401, Regression, Logistic; Odds Ratio (OR) = 0.647, 95% CI [0.427 to 0.98]
Statistical Analysis 6: Comparison: BIBR 1048 50 mg Bid vs Enoxaparin 40 mg qd; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; p = 0.2446, Regression, Logistic; Odds Ratio (OR) = 1.249, 95% CI [0.859 to 1.817]

3. Secondary Outcome: Number of Participants With Proximal DVT, PE (Pulmonary Embolism) and VTE Related Mortality
Description: Deep venous thrombosis (DVT) (proximal) as detected by routine bilateral venography on day 8 +/- 2, plus symptomatic proximal DVT confirmed by venography during the treatment period or PE confirmed by objective testing plus VTE related mortality
Time Frame: Treatment period (up to day 10)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 372 | 375 | 381 | 371 | 382
participants | 15 | 11 | 5 | 6 | 17
Statistical Analysis 1: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 225 mg Bid; BIBR 1048 225 mg bid vs. BIBR 1048 50 mg bid, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.0373, Regression, Logistic; Odds Ratio (OR) = 0.334, 95% CI [0.199 to 0.938]
Statistical Analysis 2: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 150 mg Bid; BIBR 1048 150 mg bid vs. BIBR 1048 50 mg bid, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.6659, Regression, Logistic; Odds Ratio (OR) = 0.837, 95% CI [0.374 to 1.875]
Statistical Analysis 3: Comparison: BIBR 1048 150 mg Bid vs BIBR 1048 300 mg qd; BIBR 1048 150 mg bid vs. BIBR 1048 300 mg qd, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.1882, Regression, Logistic; Odds Ratio (OR) = 0.505, 95% CI [0.183 to 1.397]
Statistical Analysis 4: Comparison: BIBR 1048 50 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 50 mg bid vs. Enoxaparin 40 mg qd, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.5566, Regression, Logistic; Odds Ratio (OR) = 0.805, 95% CI [0.39 to 1.66]
Statistical Analysis 5: Comparison: BIBR 1048 150 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 150 mg bid vs. Enoxaparin 40 mg qd, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.3253, Regression, Logistic; Odds Ratio (OR) = 0.674, 95% CI [0.307 to 1.48]
Statistical Analysis 6: Comparison: BIBR 1048 225 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 225 mg bid vs. Enoxaparin 40 mg qd, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.0114, Regression, Logistic; Odds Ratio (OR) = 0.269, 95% CI [0.097 to 0.744]

4. Secondary Outcome: Number of Participants With Proximal DVT
Description: Deep venous thrombosis (DVT) (proximal) as detected by routine bilateral venography on day 8 +/- 2, plus symptomatic proximal DVT confirmed by venography during the treatment period
Time Frame: Treatment period (up to day 8+/-2 days visit)
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Enoxaparin 40 mg qd: Enoxaparin 40 mgqd (once daily) subcutaneous injection
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 372 | 375 | 381 | 371 | 382
participants | 15 | 9 | 5 | 6 | 17
Statistical Analysis 1: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 225 mg Bid; BIBR 1048 225 mg bid vs. BIBR 1048 50 mg bid, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.036, Regression, Logistic; Odds Ratio (OR) = 0.332, 95% CI [0.118 to 0.931]
Statistical Analysis 2: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 150 mg Bid; BIBR 1048 150 mg bid vs. BIBR 1048 50 mg bid, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.3884, Regression, Logistic; Odds Ratio (OR) = 0.687, 95% CI [0.293 to 1.611]
Statistical Analysis 3: Comparison: BIBR 1048 150 mg Bid vs BIBR 1048 300 mg qd; BIBR 1048 150 mg bid vs. BIBR 1048 300 mg qd, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.3674, Regression, Logistic; Odds Ratio (OR) = 0.616, 95% CI [0.215 to 1.766]
Statistical Analysis 4: Comparison: BIBR 1048 50 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 50 mg bid vs. Enoxaparin 40 mg qd, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.5663, Regression, Logistic; Odds Ratio (OR) = 0.809, 95% CI [0.393 to 1.668]
Statistical Analysis 5: Comparison: BIBR 1048 150 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 150 mg bid vs. Enoxaparin 40 mg qd, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.1678, Regression, Logistic; Odds Ratio (OR) = 0.556, 95% CI [0.242 to 1.28]
Statistical Analysis 6: Comparison: BIBR 1048 225 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 225 mg bid vs. Enoxaparin 40 mg qd, same methodology as primary endpoint; Test type: Superiority or Other; p = 0.0113, Regression, Logistic; Odds Ratio (OR) = 0.269, 95% CI [0.097 to 0.743]

5. Primary Outcome: Number of Participants With Major Bleeding Events (MBE)
Time Frame: From approximately 14 days prior to surgery to 4-6 weeks post surgery
Population: Safety Set (SAFE) population. This included all randomised patients who were treated and who had any available data
Measure: Number; unit: participants
Groups:
- Enoxaparin 40 mg qd: Enoxaparin 40mg qd (once daily) subcutaneous injection
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 389 | 390 | 393 | 385 | 392
participants | 1 | 16 | 15 | 18 | 8
Statistical Analysis 1: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 225 mg Bid; BIBR 1048 225 mg bid vs. BIBR 1048 50 mg bid, same methodology as for primary endpoint; Test type: Superiority or Other; p = 0.0077, Regression, Logistic; Odds Ratio (OR) = 15.818, 95% CI [2.077 to 120.474]
Statistical Analysis 2: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 150 mg Bid; BIBR 1048 150 mg bid vs. BIBR 1048 50 mg bid, same methodology as for primary endpoint; Test type: Superiority or Other; p = 0.0062, Regression, Logistic; Odds Ratio (OR) = 16.907, 95% CI [2.229 to 128.238]
Statistical Analysis 3: Comparison: BIBR 1048 150 mg Bid vs BIBR 1048 300 mg qd; BIBR 1048 150 mg bid vs. BIBR 1048 300 mg qd, same methodology as for primary endpoint; Test type: Superiority or Other; p = 0.7192, Regression, Logistic; Odds Ratio (OR) = 1.136, 95% CI [0.567 to 2.276]
Statistical Analysis 4: Comparison: BIBR 1048 50 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 50 mg bid vs. Enoxaparin 40 mg qd, same methodology as for primary endpoint; Test type: Superiority or Other; p = 0.0472, Regression, Logistic; Odds Ratio (OR) = 0.121, 95% CI [0.015 to 0.974]
Statistical Analysis 5: Comparison: BIBR 1048 150 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 150 mg bid vs. Enoxaparin 40 mg qd, same methodology as for primary endpoint; Test type: Superiority or Other; p = 0.1043, Regression, Logistic; Odds Ratio (OR) = 2.049, 95% CI [0.862 to 4.868]
Statistical Analysis 6: Comparison: BIBR 1048 225 mg Bid vs Enoxaparin 40 mg qd; BIBR 1048 225 mg bid vs. Enoxaparin 40 mg qd, same methodology as for primary endpoint; Test type: Superiority or Other; p = 0.1448, Regression, Logistic; Odds Ratio (OR) = 1.917, 95% CI [0.799 to 4.597]

6. Secondary Outcome: Volume of Blood Loss
Description: Volume of blood loss was to be analysed using an analysis of variance (ANOVA), which included treatment and centre.
Time Frame: Day 1 (Day of surgery)
Population: Safety Set (SAFE) population. This included all randomised patients who were treated and who had any available data
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 389 | 390 | 393 | 385 | 392
ml | 523.3 (845.8) | 1538.4 (1474.5) | 631.4 (720.9) | 910.3 (918.3) | 945.5 (651.3)

7. Secondary Outcome: Rate of Transfusions Due to Bleedings
Description: Percentage of patients requiring transfusions due to bleeding .Rate of need of transfusion were to be analysed using a logistic regression with treatment and centre.
Time Frame: Day 1 (Day of surgery)
Population: Safety Set (SAFE) population. This included all randomised patients who were treated and who had any available data
Measure: Number; unit: Percentage of patients
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 389 | 390 | 393 | 385 | 392
Percentage of patients | 0.26 | 5.38 | 4.07 | 4.94 | 3.57
Statistical Analysis 1: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 225 mg Bid; Test type: Superiority or Other; p = 0.0063, Regression, Logistic; Odds Ratio (OR) = 16.871, 95% CI 2-sided [2.221 to 128.142]
Statistical Analysis 2: Comparison: BIBR 1048 50 mg Bid vs BIBR 1048 150 mg Bid; Test type: Superiority or Other; p = 0.0025, Regression, Logistic; Odds Ratio (OR) = 22.338, 95% CI 2-sided [2.983 to 167.268]
Statistical Analysis 3: Comparison: BIBR 1048 150 mg Bid vs BIBR 1048 300 mg qd; Test type: Superiority or Other; p = 0.7973, Regression, Logistic; Odds Ratio (OR) = 0.919, 95% CI 2-sided [0.483 to 1.750]
Statistical Analysis 4: Comparison: BIBR 1048 50 mg Bid vs Enoxaparin 40 mg qd; Test type: Superiority or Other; p = 0.0097, Regression, Logistic; Odds Ratio (OR) = 0.068, 95% CI 2-sided [0.009 to 0.522]
Statistical Analysis 5: Comparison: BIBR 1048 150 mg Bid vs Enoxaparin 40 mg qd; Test type: Superiority or Other; p = 0.2375, Regression, Logistic; Odds Ratio (OR) = 1.522, 95% CI 2-sided [0.758 to 3.058]
Statistical Analysis 6: Comparison: BIBR 1048 225 mg Bid vs Enoxaparin 40 mg qd; Test type: Superiority or Other; p = 0.7104, Regression, Logistic; Odds Ratio (OR) = 1.150, 95% CI 2-sided [0.550 to 2.403]

8. Secondary Outcome: Number of Participants With Clinically Significant, Minor or Any Bleeding Events
Description: Number of participants with Clinically Significant, minor or any bleeding events. Clinically significant bleeding events are defined as
  * Spontaneous skin haematoma larger than >25 cm²
  * Wound haematoma >100 cm²
  * Spontaneous nose bleed >5 minutes
  * Macroscopic haematurea, either spontaneous or lasting more than 24 hours if associated with an intervention
  * Spontaneous rectal bleeding (more than spot on toilet paper)
  * Gingival bleeding >5 minutes
  * Any other bleeding event considered as clinically significant by the investigator All other bleeding events that did not fulfil the criteria of MBE or clinically significant bleeding event were classified as minor bleeding events.
Time Frame: Treatment period (up to day 8+/-2 days visit)
Population: Safety Set (SAFE) population. This included all randomised patients who were treated and who had any available data
Measure: Number; unit: participants
Groups:
- BIBR 1048 150 mg Bid: Dabigatran 50 mg bid (twice daily) oral
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 389 | 390 | 393 | 385 | 392
participants
  Clinically significant bleeding events | 9 | 16 | 20 | 19 | 10
  Minor bleeding events | 18 | 31 | 38 | 37 | 25
  Any bleeding events | 26 | 61 | 65 | 62 | 43

9. Secondary Outcome: Laboratory Analyses
Description: Number of patients with possible clinically significant abnormalities, i.e. with values out of normal range.
  Normal ranges are defined as:
  Haematocrit [%]: (0.35-0.45) for women and (0.39-0.51) for men Haemoglobin [g/dL]: (11.6-15.4) for women and (13.2-17.3) for men White Blood Cell count [10^9/L]: (4-10.3) for women and (3.9-10.3) for men Platelets [10^9/L]: (145-420) for women and men Sodium [mmol/L]: (135-146) for women and men Potassium [mmol/L]: (3.5-5) for women and men Aspartate aminotransferase (AST) [U/L]: (11-37) for women and (11-39) for men Alanine aminotransferase (ALT) [U/L]: (8-43) for women and (8-45) for men Alkaline Phosphatase [U/L]: (36-118) for women and (35-123) for men Creatinine [mg/dL]: (0.57-1.06)for women and (0.72-1.3) for men Bilirubin, total [mg/dL]: (0.22-1.28) for women and men Uric acid [mg/dL]: (2.4-6.47) for women and men
Time Frame: Screening to end of treatment
Population: Safety Set (SAFE) population. This included all randomised patients who were treated and who had any available data
Measure: Number; unit: participants
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 389 | 390 | 393 | 385 | 392
participants
  Haematocrit decrease (N=325,324,339,320,340) | 16 | 15 | 14 | 14 | 22
  Haemoglobin decrease (N=325,324,339,320,340) | 122 | 129 | 148 | 129 | 142
  White blood cell ct. decr.(N=325,324,339,320,340) | 0 | 0 | 2 | 1 | 0
  Platelets decrease (N=325,324,339,320,340) | 0 | 0 | 0 | 0 | 1
  Platelets increase (N=325,324,339,320,340) | 0 | 1 | 1 | 0 | 0
  Sodium decrease (N=340,334,344,327,352) | 0 | 2 | 0 | 1 | 0
  Potassium decrease (N=340,334,344,326,352) | 0 | 0 | 1 | 0 | 2
  Potassium increase (N=340,334,344,326,352) | 0 | 2 | 1 | 2 | 1
  AST increase (N=340,334,344,327,352) | 1 | 0 | 2 | 3 | 9
  ALT increase (N=340,334,344,327,352) | 6 | 5 | 3 | 8 | 20
  Alkaline phosphatase incr. (N=340,334,344,327,352) | 1 | 2 | 0 | 0 | 3
  Creatinine increase (N=340,334,344,327,352) | 0 | 2 | 0 | 1 | 1
  Bilirubin, total increase (N=340,334,344,327,352) | 0 | 0 | 0 | 1 | 0
  Uric Acid increase (N=340,334,344,327,352) | 3 | 4 | 4 | 2 | 3

10. Secondary Outcome: Plasma Concentration (Cmax) of Dabigatran
Description: Maximum plasma concentration of Dabigatran (at steady-state) and Pre-dose plasma concentrations at steady state.
  Cmax represents the maximum concentration of Dabigatran in plasma. Cmax,ss represents the maximum concentration of Dabigatran in plasma at steady state.
  Cpre,ss represents pre-dose concentration of Dabigatran in plasma at steady state
Time Frame: Day 1 to end of treatment
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 365 | 358 | 365 | 351 | 0
ng/mL
  Cmax (N=88, 83, 84, 96, 0) | 24.5 (115) | 60.5 (97.3) | 79.9 (94.7) | 132 (81.6) |
  Cmax at steady-state (N=87, 74, 79, 85, 0) | 48.0 (64.6) | 165 (63.6) | 257 (62.7) | 271 (75.2) |
  Cpre at steady-state | 19.6 (70.7) | 70.3 (87.3) | 113 (80.9) | 38.0 (85.9) |

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve During a Dosing Interval
Description: Area under the plasma concentration-time curve during a dosing interval (at steady-state). The AUC0-12h (for b.i.d. treatment regimens) and AUC0-24h (300 mg q.d.) after the first dose on day of surgery calculated by extrapolation using the elimination rate constant, reported only if the extrapolated fraction of AUC was less than 30 % of the total AUC.
Time Frame: up to day 8+/-2 days visit
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Number analyzed (Participants) | 69 | 54 | 62 | 76 | 0
ng*h/mL
  AUC during a dosing interval (N=13,12,21,72,0) | 229 (88.1) | 636 (56.2) | 605 (91.6) | 1610 (82.5) |
  AUC during a dosing interval at steady-state | 350 (66.8) | 1250 (64.8) | 1910 (64.9) | 2450 (76.1) |

ADVERSE EVENTS:
Time Frame: 14 days +/- 2 days
Description: Time frame is from first dose of randomised treatment up to the end of treatment including 6 days after last intake.
Arm/Group | BIBR 1048 50 mg Bid | BIBR 1048 150 mg Bid | BIBR 1048 225 mg Bid | BIBR 1048 300 mg qd | Enoxaparin 40 mg qd
Serious Adverse Events (participants affected / at risk) | 25/389 | 29/390 | 21/393 | 33/385 | 31/392
Other Adverse Events (participants affected / at risk) | 242/389 | 267/390 | 256/393 | 267/385 | 258/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIBR 1048 50 mg Bid (N=389) | BIBR 1048 150 mg Bid (N=390) | BIBR 1048 225 mg Bid (N=393) | BIBR 1048 300 mg qd (N=385) | Enoxaparin 40 mg qd (N=392)
Haemolytic anaemia NOS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Leukopenia NOS (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Bradycardia NOS (Cardiac disorders) | 0 | 1 | 0 | 1 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac disorder NOS (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 0 | 1 | 0
Fall (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Hyperpyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 1 | 0 | 0
Inflammation localised (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema lower limb (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0
Rigors (General disorders) | 0 | 0 | 0 | 0 | 1
Arthritis infective NOS (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Bronchopneumonia NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cystitis NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis NOS (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Implant infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Meningitis NOS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia NOS (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Post-operative wound infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Wound infection NEC (Infections and infestations) | 1 | 1 | 3 | 3 | 3
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femur fracture NOS (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 1
Haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Intraoperative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Joint dislocation NEC (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 3 | 1
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Joint ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural drainage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 3 | 1
Post procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Postoperative haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0
Blood alkaline phosphatase NOS increased (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Bone disorder NOS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Rheumatoid arthritis aggravated (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Colon cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Colon neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Lung neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Epilepsy NOS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic stroke NOS (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral neuropathy NOS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Radiculitis NOS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal failure aggravated (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Face oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Arterial haemorrhage NOS (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Deep venous thrombosis NOS (Vascular disorders) | 1 | 0 | 0 | 1 | 3
Haematoma NOS (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhage NOS (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension NOS (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Vascular disorders) | 1 | 3 | 0 | 0 | 0
Venous thrombosis deep limb (Vascular disorders) | 5 | 1 | 1 | 1 | 2
Wound haemorrhage (Vascular disorders) | 0 | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIBR 1048 50 mg Bid (N=389) | BIBR 1048 150 mg Bid (N=390) | BIBR 1048 225 mg Bid (N=393) | BIBR 1048 300 mg qd (N=385) | Enoxaparin 40 mg qd (N=392)
Anaemia NOS (Blood and lymphatic system disorders) | 23 | 26 | 27 | 22 | 18
Constipation (Gastrointestinal disorders) | 33 | 38 | 34 | 46 | 34
Nausea (Gastrointestinal disorders) | 84 | 105 | 92 | 105 | 111
Vomiting NOS (Gastrointestinal disorders) | 76 | 77 | 75 | 76 | 66
Pyrexia (General disorders) | 33 | 30 | 36 | 35 | 32
Post procedural drainage (Injury, poisoning and procedural complications) | 12 | 16 | 23 | 18 | 8
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 6 | 14 | 6 | 18 | 20
Wound secretion (Injury, poisoning and procedural complications) | 15 | 21 | 16 | 17 | 6
Haemoglobin decreased (Investigations) | 13 | 18 | 21 | 15 | 21
Headache NOS (Nervous system disorders) | 19 | 15 | 16 | 10 | 20
Insomnia (Psychiatric disorders) | 59 | 45 | 52 | 59 | 51
Haematoma NOS (Vascular disorders) | 10 | 17 | 21 | 14 | 5
Hypotension NOS (Vascular disorders) | 19 | 25 | 21 | 21 | 20
Venous thrombosis deep limb (Vascular disorders) | 33 | 12 | 13 | 12 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.